CLINICAL TRIAL: NCT01509690
Title: Impact of a Multidisciplinary Intensive Management Clinic on Clinical, Patient-Reported and Economic Outcomes in Multi-Ethnic Asian Incident Hemodialysis Patients
Brief Title: Impact of a Multidisciplinary Intensive Management Clinic on Outcomes in Multi-Ethnic Asian Incident Hemodialysis Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Priscilla How, Pharm.D., BCPS, Assistant Professor, National University of Singapore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: DSRB Domain E/2011/1772
Record Dates: First submitted 2012-01-06; First posted 2012-01-13 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Stage 5 Chronic Kidney Disease
Keywords: Incident; Hemodialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Multidisciplinary, intensive and collaborative care — No specific study drugs, devices or procedures are involved.
  Subjects will be seen in a multidisciplinary, intensive management clinic involving a renal physician, a clinical pharmacist trained in renal pharmacotherapy and a renal coordinator. The main aim of this clinic is to provide multidisciplinary, intensive and consistent care in the first 3 to 4 months after HD initiation to streamline the management of the patients. Specific objectives of this clinic include providing patients with educational materials and information to enable a better understanding of their disease process, providing uniform anemia and renal bone disease management, increasing permanent HD access [arteriovenous (AV) fistula or graft] placement, increasing transplant referrals, providing suitable vaccinations to all patients, as well as reducing hospitalizations for fluid overload, uncontrolled hypertension and anemia-related complications.
  Other Names: No specific study drugs, devices or procedures are involved

SUMMARY:
Patients with end-stage renal disease are most vulnerable in the early months following hemodialysis (HD) initiation. Data from the United States Renal Data System and Singapore Renal Registry showed high mortality rates in the first 3-12 months of dialysis. Comprehensive multidisciplinary intervention programs implemented in the initial 3-4 months of dialysis showed reduction in mortality and morbidity in incident dialysis patients in the United States.

Based on these models, the Hemodialysis Initiation and Transition (HIT) Clinic involving a renal physician, clinical pharmacist and coordinator was set up. The main aim of the clinic is to provide multidisciplinary, intensive and consistent care to patients in the first 3 to 4 months after HD initiation to focus on and streamline the management of dialysis issues and complications. These interventions would help patients achieve goal therapeutic targets, as well as reduce hospitalization rates and mortality, thereby improving their clinical outcomes and self-reported quality of life, and could result in economic and cost savings for the patients and healthcare system. The purpose of this study is to determine if the multidisciplinary, intensive and collaborative management of our multiethnic Asian patients newly-initiated on HD improves laboratory, clinical, economic and patient-reported outcomes.

Adult incident HD patients from NUH will be randomized to the HIT clinic or to conventional management. Information on demographics, medical/medication histories, laboratory data (dialysis adequacy, iron-deficiency anemia, mineral/bone disorder, malnutrition and diabetes), hospitalizations, deaths and medical costs will be obtained and compared between the 2 groups. Patient-reported outcomes will be measured using the Kidney Disease Quality of Life-Short Form, EuroQol 5 Dimensions, Family Functioning Measure, Oslo-3 Social Support Scale and Health Services Utilization questionnaires. Data collection will take place at baseline, 3 to 4 months and 12 months after the first visit, with a total study duration and follow-up period of 1 year.

ELIGIBILITY:
Inclusion Criteria:

* all patients who are newly-initiated on HD and who meet the following criteria will be included in the study:
* male or female 21 years of age or older with stage 5 CKD (eGFR < 15 ml/min/1.73m2)
* newly-initiated on HD within the past 4-8 weeks of being seen in the NUH outpatient renal clinic

Exclusion Criteria:

* transient HD patients
* patients with poor cognitive function or are not able to complete the PRO questionnaires.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)

PRIMARY OUTCOMES:
Clinical (mortality and morbidity) | One year
  Mortality and morbidity (hospitalization from uncontrolled hypertension, anemia and fluid overload)

SECONDARY OUTCOMES:
Laboratory outcomes | One year
  Lab results
Economic outcomes | One year
  Direct and indirect medical costs
Patient-reported outcomes | One-year
  KDQOL and other social support questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla P How, Pharm.D., BCPS, Principal Investigator — National University of Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore